CLINICAL TRIAL: NCT01931852
Title: Cardiac Magnetic Resonance Imaging Strategy for the Management of Patients With Acute Chest Pain and Detectable to Elevated Troponin
Acronym: CMR-IMPACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: IRB00022322; 1R01HL118263-01A1 (NIH)
Record Dates: First submitted 2013-08-26; First posted 2013-08-29 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2020-07

CONDITIONS: Acute Coronary Syndrome; Chest Pain
Keywords: Acute Coronary Syndrome; Chest pain; Cardiac MRI; Risk Stratification; Emergency Department; Elevated Troponin; Troponin; Non-ST Elevation Myocardial Infarction
MeSH Terms: conditions — Acute Coronary Syndrome; Chest Pain; Emergencies; Non-ST Elevated Myocardial Infarction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CMR-guided care (Experimental): Participants in this group will receive a cardiac MRI
  Interventions: Procedure: Cardiac MRI
- Invasive-based guideline-adherent care (Active Comparator): Participants will receive care adherent with current ACC/AHA guideline recommendations. ( ACC/AHA Guideline adherent care )
  Interventions: Other: ACC/AHA Guideline adherent care

INTERVENTIONS:
Procedure: Cardiac MRI — Participants in the CMR-guided care group will receive a cardiac MRI.
  Other Names: CMR; Cardiac Magnetic Resonance Imaging
  Arms: CMR-guided care
Other: ACC/AHA Guideline adherent care — Participants in the invasive-based guideline-adherent care group will receive care adherent with current American College of Cardiology / American Heart Association (ACC/AHA) guideline recommendations. ( ACC/AHA Guideline adherent care )
  Arms: Invasive-based guideline-adherent care

SUMMARY:
The broad, long-term objective is to improve outcomes by optimizing healthcare delivery processes for patients with detectable to elevated serum troponin. This clinical trial involving emergency department (ED) patients with intermediate to high-risk chest pain and detectable to minimally elevated serum troponin within 6 hours of evaluation.

DETAILED DESCRIPTION:
In the evaluation of patients with possible acute coronary syndrome, serum troponin measurement is a critical determinant of myocardial necrosis. The recent implementation of high-sensitivity troponin assays allows detection of lower levels of serum troponin than possible with less sensitive predecessors. As a result, 30% more patients are diagnosed with myocardial injury but the optimal management of these patients is unclear. Guidelines from the American Heart Association and American College of Cardiology recommend an invasive management strategy (Class 1a) but acknowledge that data supporting an invasive strategy were based on less sensitive troponin assays than those available today. Clinical trials of an invasive strategy in patients with detectable to minimally elevated troponin values demonstrate conflicting results. Observational data suggest aggressive medical therapy rather than increased use of revascularization drives improved outcomes in these patients. Meanwhile, these patients with minimally elevated serum troponin values have experienced a near doubling in the rate of invasive angiography. In short, it is uncertain whether patients with detectable to minimally elevated troponin results benefit from current invasive-based care strategies. As an alternative, cardiac magnetic resonance (CMR) imaging is highly accurate for detecting significant coronary disease and the need for coronary revascularization.

Objectives: The broad, long-term objective is to improve outcomes by optimizing healthcare delivery processes for patients with detectable to elevated serum troponin. To achieve this goal, we propose a clinical trial (n=312) involving emergency department patients with intermediate to high-risk chest pain and detectable to minimally elevated serum troponin within 6 hours of evaluation.

Methods: Participants will be randomized to one of two care strategies: a) invasive-based guideline-adherent strategy, or b) CMR-guided. Outcomes will be assessed over an average of 2.3 years. The specific aims of this proposal are 1) Test whether a CMR-guided strategy (versus invasive-based guideline-adherent strategy) reduces the composite of death, nonfatal myocardial infarction, and cardiac-related hospital readmission over the study duration, and 2) Test whether a CMR-guided strategy (versus invasive-based guideline-adherent strategy) reduces invasive angiography, coronary revascularization, recurrent cardiac testing, and cardiac-related emergency department visits.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 21 years of age at the time of enrollment
* Symptoms consistent with acute coronary syndrome
* At least 1 troponin > lower limit of detection and ≤1.0 ng/ml within 6 hours of the initial evaluation

Exclusion Criteria:

* Any troponin >1.0 ng/ml at the time of consent
* New ST-segment elevation (≥ 1 mV) or depression (≥ 2 mV)
* Hemodynamic instability (symptomatic systolic BP <90 mmHg, dysrhythmia)
* Ongoing, unrelieved symptoms thought to represent cardiac ischemia and requiring immediate cardiac catheterization
* Known severe multi-vessel CAD previously determined to be not amendable to mechanical intervention
* Coronary revascularization in the past 6 months
* Contra-indications to magnetic resonance imaging Examples: Unable to lie flat, pacemaker, defibrillator, cerebral aneurysm clips, metallic ocular foreign body, implanted devices, severe claustrophobia, pregnancy
* Life expectancy less than 12 months
* Increased risk for nephrogenic systemic fibrosis i. Creatinine clearance < 30 ml/min at the time of enrollment ii. clinical concern for acute kidney injury and/or acute renal failure* iii. Hepato-renal syndrome or chronic liver disease with a creatinine clearance of <60 ml/min at the time of enrollment iv. History of liver, heart, or kidney transplant

  * This may be manifested by a recent or concurrent rise in serum creatinine, or a reduction in baseline creatinine clearance.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 312 (Actual)
Dates: Start 2013-09 (Actual); Primary Completion 2020-07-29 (Actual); Study Completion 2020-10-02 (Actual)

PRIMARY OUTCOMES:
Reduction in composite death, nonfatal myocardial infarction (MI), cardiac-related hospital readmissions, and cardiac-related Emergency Department (ED) visits. | 5 years
  Test whether a CMR-guided strategy (versus invasive-based guideline-adherent strategy) reduces the composite of death, nonfatal MI, cardiac-related hospital readmission, and cardiac-related ED visits over time.

SECONDARY OUTCOMES:
Reduction in invasive angiography. | 5 years
  Test whether a CMR-guided strategy (versus invasive-based guideline-adherent strategy) reduces invasive angiography.
Reduction in coronary revascularization. | 5 years
  Test whether a CMR-guided strategy (versus invasive-based guideline-adherent strategy) reduces coronary revascularization.
Reduction in recurrent cardiac testing. | 5 years
  Test whether a CMR-guided strategy (versus invasive-based guideline-adherent strategy) reduces recurrent cardiac testing.

CONTACTS AND LOCATIONS:
Overall Officials: Chadwick Miller, MD, MS, Principal Investigator — WFBMC
Locations (4):
- United States (4):
  - William Beaumont Hospital, Royal Oak, Michigan
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Wake Forest Baptist Medical Center, Winston-Salem, North Carolina
  - The Ohio State University Wexner Medical Center, Columbus, Ohio

REFERENCES:
- [Background] Pitts SR, Niska RW, Xu J, Burt CW. National Hospital Ambulatory Medical Care Survey: 2006 emergency department summary. Natl Health Stat Report. 2008 Aug 6;(7):1-38. PMID 18958996
- [Background] Christenson J, Innes G, McKnight D, Thompson CR, Wong H, Yu E, Boychuk B, Grafstein E, Rosenberg F, Gin K, Anis A, Singer J. A clinical prediction rule for early discharge of patients with chest pain. Ann Emerg Med. 2006 Jan;47(1):1-10. doi: 10.1016/j.annemergmed.2005.08.007. Epub 2005 Oct 19. PMID 16387209
- [Background] Wright RS, Anderson JL, Adams CD, Bridges CR, Casey DE Jr, Ettinger SM, Fesmire FM, Ganiats TG, Jneid H, Lincoff AM, Peterson ED, Philippides GJ, Theroux P, Wenger NK, Zidar JP, Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS. 2011 ACCF/AHA focused update of the Guidelines for the Management of Patients with Unstable Angina/Non-ST-Elevation Myocardial Infarction (updating the 2007 guideline): a report of the American College of Cardiology Foundation/American Heart Association Task Force on Practice Guidelines developed in collaboration with the American College of Emergency Physicians, Society for Cardiovascular Angiography and Interventions, and Society of Thoracic Surgeons. J Am Coll Cardiol. 2011 May 10;57(19):1920-59. doi: 10.1016/j.jacc.2011.02.009. Epub 2011 Mar 28. No abstract available. PMID 21450428
- [Background] Tatum JL, Jesse RL, Kontos MC, Nicholson CS, Schmidt KL, Roberts CS, Ornato JP. Comprehensive strategy for the evaluation and triage of the chest pain patient. Ann Emerg Med. 1997 Jan;29(1):116-25. doi: 10.1016/s0196-0644(97)70317-2. PMID 8998090
- [Background] Hoffmann U, Nagurney JT, Moselewski F, Pena A, Ferencik M, Chae CU, Cury RC, Butler J, Abbara S, Brown DF, Manini A, Nichols JH, Achenbach S, Brady TJ. Coronary multidetector computed tomography in the assessment of patients with acute chest pain. Circulation. 2006 Nov 21;114(21):2251-60. doi: 10.1161/CIRCULATIONAHA.106.634808. Epub 2006 Oct 30. PMID 17075011
- [Background] Gomberg-Maitland M, Murphy SA, Moliterno DJ, Cannon CP. Are we appropriately triaging patients with unstable angina? Am Heart J. 2005 Apr;149(4):613-8. doi: 10.1016/j.ahj.2004.09.035. PMID 15990742
- [Background] Stowers SA, Eisenstein EL, Th Wackers FJ, Berman DS, Blackshear JL, Jones AD Jr, Szymanski TJ Jr, Lam LC, Simons TA, Natale D, Paige KA, Wagner GS. An economic analysis of an aggressive diagnostic strategy with single photon emission computed tomography myocardial perfusion imaging and early exercise stress testing in emergency department patients who present with chest pain but nondiagnostic electrocardiograms: results from a randomized trial. Ann Emerg Med. 2000 Jan;35(1):17-25. doi: 10.1016/S0196-0644(00)70100-4. PMID 10613936
- [Background] Goldstein JA, Gallagher MJ, O'Neill WW, Ross MA, O'Neil BJ, Raff GL. A randomized controlled trial of multi-slice coronary computed tomography for evaluation of acute chest pain. J Am Coll Cardiol. 2007 Feb 27;49(8):863-71. doi: 10.1016/j.jacc.2006.08.064. Epub 2007 Feb 12. PMID 17320744
- [Background] Heller GV, Stowers SA, Hendel RC, Herman SD, Daher E, Ahlberg AW, Baron JM, Mendes de Leon CF, Rizzo JA, Wackers FJ. Clinical value of acute rest technetium-99m tetrofosmin tomographic myocardial perfusion imaging in patients with acute chest pain and nondiagnostic electrocardiograms. J Am Coll Cardiol. 1998 Apr;31(5):1011-7. doi: 10.1016/s0735-1097(98)00057-6. PMID 9562001
- [Background] Farkouh ME, Smars PA, Reeder GS, Zinsmeister AR, Evans RW, Meloy TD, Kopecky SL, Allen M, Allison TG, Gibbons RJ, Gabriel SE. A clinical trial of a chest-pain observation unit for patients with unstable angina. Chest Pain Evaluation in the Emergency Room (CHEER) Investigators. N Engl J Med. 1998 Dec 24;339(26):1882-8. doi: 10.1056/NEJM199812243392603. PMID 9862943
- [Background] Body R, Carley S, McDowell G, Jaffe AS, France M, Cruickshank K, Wibberley C, Nuttall M, Mackway-Jones K. Rapid exclusion of acute myocardial infarction in patients with undetectable troponin using a high-sensitivity assay. J Am Coll Cardiol. 2011 Sep 20;58(13):1332-9. doi: 10.1016/j.jacc.2011.06.026. PMID 21920261
- [Background] Mills NL, Churchhouse AM, Lee KK, Anand A, Gamble D, Shah AS, Paterson E, MacLeod M, Graham C, Walker S, Denvir MA, Fox KA, Newby DE. Implementation of a sensitive troponin I assay and risk of recurrent myocardial infarction and death in patients with suspected acute coronary syndrome. JAMA. 2011 Mar 23;305(12):1210-6. doi: 10.1001/jama.2011.338. PMID 21427373
- [Background] Mehta SR, Cannon CP, Fox KA, Wallentin L, Boden WE, Spacek R, Widimsky P, McCullough PA, Hunt D, Braunwald E, Yusuf S. Routine vs selective invasive strategies in patients with acute coronary syndromes: a collaborative meta-analysis of randomized trials. JAMA. 2005 Jun 15;293(23):2908-17. doi: 10.1001/jama.293.23.2908. PMID 15956636
- [Background] Cannon CP, Weintraub WS, Demopoulos LA, Vicari R, Frey MJ, Lakkis N, Neumann FJ, Robertson DH, DeLucca PT, DiBattiste PM, Gibson CM, Braunwald E; TACTICS (Treat Angina with Aggrastat and Determine Cost of Therapy with an Invasive or Conservative Strategy)--Thrombolysis in Myocardial Infarction 18 Investigators. Comparison of early invasive and conservative strategies in patients with unstable coronary syndromes treated with the glycoprotein IIb/IIIa inhibitor tirofiban. N Engl J Med. 2001 Jun 21;344(25):1879-87. doi: 10.1056/NEJM200106213442501. PMID 11419424
- [Background] Qayyum R, Khalid MR, Adomaityte J, Papadakos SP, Messineo FC. Systematic review: comparing routine and selective invasive strategies for the acute coronary syndrome. Ann Intern Med. 2008 Feb 5;148(3):186-96. doi: 10.7326/0003-4819-148-3-200802050-00005. PMID 18252682
- [Background] McCullough PA, O'Neill WW, Graham M, Stomel RJ, Rogers F, David S, Farhat A, Kazlauskaite R, Al-Zagoum M, Grines CL. A prospective randomized trial of triage angiography in acute coronary syndromes ineligible for thrombolytic therapy. Results of the medicine versus angiography in thrombolytic exclusion (MATE) trial. J Am Coll Cardiol. 1998 Sep;32(3):596-605. doi: 10.1016/s0735-1097(98)00284-8. PMID 9741499
- [Background] Fox KA, Poole-Wilson P, Clayton TC, Henderson RA, Shaw TR, Wheatley DJ, Knight R, Pocock SJ. 5-year outcome of an interventional strategy in non-ST-elevation acute coronary syndrome: the British Heart Foundation RITA 3 randomised trial. Lancet. 2005 Sep 10-16;366(9489):914-20. doi: 10.1016/S0140-6736(05)67222-4. PMID 16154018
- [Background] Michalis LK, Stroumbis CS, Pappas K, Sourla E, Niokou D, Goudevenos JA, Siogas C, Sideris DA. Treatment of refractory unstable angina in geographically isolated areas without cardiac surgery. Invasive versus conservative strategy (TRUCS study). Eur Heart J. 2000 Dec;21(23):1954-9. doi: 10.1053/euhj.2000.2397. PMID 11071801
- [Background] Lagerqvist B, Husted S, Kontny F, Stahle E, Swahn E, Wallentin L; Fast Revascularisation during InStability in Coronary artery disease (FRISC-II) Investigators. 5-year outcomes in the FRISC-II randomised trial of an invasive versus a non-invasive strategy in non-ST-elevation acute coronary syndrome: a follow-up study. Lancet. 2006 Sep 16;368(9540):998-1004. doi: 10.1016/S0140-6736(06)69416-6. PMID 16980115
- [Background] Hirsch A, Windhausen F, Tijssen JG, Verheugt FW, Cornel JH, de Winter RJ; Invasive versus Conservative Treatment in Unstable coronary Syndromes (ICTUS) investigators. Long-term outcome after an early invasive versus selective invasive treatment strategy in patients with non-ST-elevation acute coronary syndrome and elevated cardiac troponin T (the ICTUS trial): a follow-up study. Lancet. 2007 Mar 10;369(9564):827-835. doi: 10.1016/S0140-6736(07)60410-3. PMID 17350451
- [Background] Boden WE, O'Rourke RA, Crawford MH, Blaustein AS, Deedwania PC, Zoble RG, Wexler LF, Kleiger RE, Pepine CJ, Ferry DR, Chow BK, Lavori PW. Outcomes in patients with acute non-Q-wave myocardial infarction randomly assigned to an invasive as compared with a conservative management strategy. Veterans Affairs Non-Q-Wave Infarction Strategies in Hospital (VANQWISH) Trial Investigators. N Engl J Med. 1998 Jun 18;338(25):1785-92. doi: 10.1056/NEJM199806183382501. PMID 9632444
- [Background] Spacek R, Widimsky P, Straka Z, Jiresova E, Dvorak J, Polasek R, Karel I, Jirmar R, Lisa L, Budesinsky T, Malek F, Stanka P. Value of first day angiography/angioplasty in evolving Non-ST segment elevation myocardial infarction: an open multicenter randomized trial. The VINO Study. Eur Heart J. 2002 Feb;23(3):230-8. doi: 10.1053/euhj.2001.2735. PMID 11792138
- [Background] Plein S, Greenwood JP, Ridgway JP, Cranny G, Ball SG, Sivananthan MU. Assessment of non-ST-segment elevation acute coronary syndromes with cardiac magnetic resonance imaging. J Am Coll Cardiol. 2004 Dec 7;44(11):2173-81. doi: 10.1016/j.jacc.2004.08.056. PMID 15582315
- [Background] Raman SV, Simonetti OP, Winner MW 3rd, Dickerson JA, He X, Mazzaferri EL Jr, Ambrosio G. Cardiac magnetic resonance with edema imaging identifies myocardium at risk and predicts worse outcome in patients with non-ST-segment elevation acute coronary syndrome. J Am Coll Cardiol. 2010 Jun 1;55(22):2480-8. doi: 10.1016/j.jacc.2010.01.047. PMID 20510215
- [Background] Miller CD, Hwang W, Case D, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Hundley WG. Stress CMR imaging observation unit in the emergency department reduces 1-year medical care costs in patients with acute chest pain: a randomized study for comparison with inpatient care. JACC Cardiovasc Imaging. 2011 Aug;4(8):862-70. doi: 10.1016/j.jcmg.2011.04.016. PMID 21835378
- [Background] Anderson JL, Adams CD, Antman EM, Bridges CR, Califf RM, Casey DE Jr, Chavey WE 2nd, Fesmire FM, Hochman JS, Levin TN, Lincoff AM, Peterson ED, Theroux P, Wenger NK, Wright RS, Smith SC Jr, Jacobs AK, Halperin JL, Hunt SA, Krumholz HM, Kushner FG, Lytle BW, Nishimura R, Ornato JP, Page RL, Riegel B; American College of Cardiology; American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction); American College of Emergency Physicians; Society for Cardiovascular Angiography and Interventions; Society of Thoracic Surgeons; American Association of Cardiovascular and Pulmonary Rehabilitation; Society for Academic Emergency Medicine. ACC/AHA 2007 guidelines for the management of patients with unstable angina/non ST-elevation myocardial infarction: a report of the American College of Cardiology/American Heart Association Task Force on Practice Guidelines (Writing Committee to Revise the 2002 Guidelines for the Management of Patients With Unstable Angina/Non ST-Elevation Myocardial Infarction): developed in collaboration with the American College of Emergency Physicians, the Society for Cardiovascular Angiography and Interventions, and the Society of Thoracic Surgeons: endorsed by the American Association of Cardiovascular and Pulmonary Rehabilitation and the Society for Academic Emergency Medicine. Circulation. 2007 Aug 14;116(7):e148-304. doi: 10.1161/CIRCULATIONAHA.107.181940. Epub 2007 Aug 6. No abstract available. PMID 17679616
- [Background] Hoffmann U, Bamberg F, Chae CU, Nichols JH, Rogers IS, Seneviratne SK, Truong QA, Cury RC, Abbara S, Shapiro MD, Moloo J, Butler J, Ferencik M, Lee H, Jang IK, Parry BA, Brown DF, Udelson JE, Achenbach S, Brady TJ, Nagurney JT. Coronary computed tomography angiography for early triage of patients with acute chest pain: the ROMICAT (Rule Out Myocardial Infarction using Computer Assisted Tomography) trial. J Am Coll Cardiol. 2009 May 5;53(18):1642-50. doi: 10.1016/j.jacc.2009.01.052. PMID 19406338
- [Background] Hollander JE, Chang AM, Shofer FS, McCusker CM, Baxt WG, Litt HI. Coronary computed tomographic angiography for rapid discharge of low-risk patients with potential acute coronary syndromes. Ann Emerg Med. 2009 Mar;53(3):295-304. doi: 10.1016/j.annemergmed.2008.09.025. Epub 2008 Nov 8. PMID 18996620
- [Background] Mahler SA, Hiestand BC, Goff DC Jr, Hoekstra JW, Miller CD. Can the HEART score safely reduce stress testing and cardiac imaging in patients at low risk for major adverse cardiac events? Crit Pathw Cardiol. 2011 Sep;10(3):128-33. doi: 10.1097/HPC.0b013e3182315a85. PMID 21989033
- [Background] Arbab-Zadeh A, Miller JM, Rochitte CE, Dewey M, Niinuma H, Gottlieb I, Paul N, Clouse ME, Shapiro EP, Hoe J, Lardo AC, Bush DE, de Roos A, Cox C, Brinker J, Lima JA. Diagnostic accuracy of computed tomography coronary angiography according to pre-test probability of coronary artery disease and severity of coronary arterial calcification. The CORE-64 (Coronary Artery Evaluation Using 64-Row Multidetector Computed Tomography Angiography) International Multicenter Study. J Am Coll Cardiol. 2012 Jan 24;59(4):379-87. doi: 10.1016/j.jacc.2011.06.079. PMID 22261160
- [Background] Hundley WG. The use of cardiovascular magnetic resonance to identify adverse cardiac prognosis: an important step in reducing image-related heath care expenditures. J Am Coll Cardiol. 2010 Oct 5;56(15):1244-6. doi: 10.1016/j.jacc.2010.07.011. No abstract available. PMID 20883931
- [Background] Miller CD, Hwang W, Hoekstra JW, Case D, Lefebvre C, Blumstein H, Hiestand B, Diercks DB, Hamilton CA, Harper EN, Hundley WG. Stress cardiac magnetic resonance imaging with observation unit care reduces cost for patients with emergent chest pain: a randomized trial. Ann Emerg Med. 2010 Sep;56(3):209-219.e2. doi: 10.1016/j.annemergmed.2010.04.009. Epub 2010 May 31. PMID 20554078
- [Background] Miller CD, Hoekstra JW, Lefebvre C, Blumstein H, Hamilton CA, Harper EN, Mahler S, Diercks DB, Neiberg R, Hundley WG. Provider-directed imaging stress testing reduces health care expenditures in lower-risk chest pain patients presenting to the emergency department. Circ Cardiovasc Imaging. 2012 Jan;5(1):111-8. doi: 10.1161/CIRCIMAGING.111.965293. Epub 2011 Nov 29. PMID 22128195
- [Background] Abdel-Aty H, Zagrosek A, Schulz-Menger J, Taylor AJ, Messroghli D, Kumar A, Gross M, Dietz R, Friedrich MG. Delayed enhancement and T2-weighted cardiovascular magnetic resonance imaging differentiate acute from chronic myocardial infarction. Circulation. 2004 May 25;109(20):2411-6. doi: 10.1161/01.CIR.0000127428.10985.C6. Epub 2004 May 3. PMID 15123531
- [Background] Cury RC, Shash K, Nagurney JT, Rosito G, Shapiro MD, Nomura CH, Abbara S, Bamberg F, Ferencik M, Schmidt EJ, Brown DF, Hoffmann U, Brady TJ. Cardiac magnetic resonance with T2-weighted imaging improves detection of patients with acute coronary syndrome in the emergency department. Circulation. 2008 Aug 19;118(8):837-44. doi: 10.1161/CIRCULATIONAHA.107.740597. Epub 2008 Aug 4. PMID 18678772
- [Background] de Winter RJ, Windhausen F, Cornel JH, Dunselman PH, Janus CL, Bendermacher PE, Michels HR, Sanders GT, Tijssen JG, Verheugt FW; Invasive versus Conservative Treatment in Unstable Coronary Syndromes (ICTUS) Investigators. Early invasive versus selectively invasive management for acute coronary syndromes. N Engl J Med. 2005 Sep 15;353(11):1095-104. doi: 10.1056/NEJMoa044259. PMID 16162880
- [Background] Menzin J, Wygant G, Hauch O, Jackel J, Friedman M. One-year costs of ischemic heart disease among patients with acute coronary syndromes: findings from a multi-employer claims database. Curr Med Res Opin. 2008 Feb;24(2):461-8. doi: 10.1185/030079908x261096. PMID 18194592
- [Background] Curtis JP, Schreiner G, Wang Y, Chen J, Spertus JA, Rumsfeld JS, Brindis RG, Krumholz HM. All-cause readmission and repeat revascularization after percutaneous coronary intervention in a cohort of medicare patients. J Am Coll Cardiol. 2009 Sep 1;54(10):903-7. doi: 10.1016/j.jacc.2009.04.076. PMID 19712799
- [Background] Medicare Payment Advisory Commission.
- [Background] National Hospital Ambulatory Medical Care Survey: 2008 Emergency Department Summary Tables. Available at: http://www.cdc.gov/nchs/data/ahcd/nhamcs_emergency/nhamcsed2008.pdf (accessed 4/11/2011).
- [Background] Bayley MD, Schwartz JS, Shofer FS, Weiner M, Sites FD, Traber KB, Hollander JE. The financial burden of emergency department congestion and hospital crowding for chest pain patients awaiting admission. Ann Emerg Med. 2005 Feb;45(2):110-7. doi: 10.1016/j.annemergmed.2004.09.010. PMID 15671965
- [Background] Diercks DB, Roe MT, Chen AY, Peacock WF, Kirk JD, Pollack CV Jr, Gibler WB, Smith SC Jr, Ohman M, Peterson ED. Prolonged emergency department stays of non-ST-segment-elevation myocardial infarction patients are associated with worse adherence to the American College of Cardiology/American Heart Association guidelines for management and increased adverse events. Ann Emerg Med. 2007 Nov;50(5):489-96. doi: 10.1016/j.annemergmed.2007.03.033. Epub 2007 Jun 20. PMID 17583379
- [Background] Miro O, Antonio MT, Jimenez S, De Dios A, Sanchez M, Borras A, Milla J. Decreased health care quality associated with emergency department overcrowding. Eur J Emerg Med. 1999 Jun;6(2):105-7. doi: 10.1097/00063110-199906000-00003. PMID 10461551
- [Background] Sprivulis PC, Da Silva JA, Jacobs IG, Frazer AR, Jelinek GA. The association between hospital overcrowding and mortality among patients admitted via Western Australian emergency departments. Med J Aust. 2006 Mar 6;184(5):208-12. doi: 10.5694/j.1326-5377.2006.tb00416.x. PMID 16515429
- [Background] Gilligan P, Winder S, Singh I, Gupta V, Kelly PO, Hegarty D. The Boarders in the Emergency Department (BED) study. Emerg Med J. 2008 May;25(5):265-9. doi: 10.1136/emj.2007.048173. PMID 18434458
- [Background] Richardson DB. Increase in patient mortality at 10 days associated with emergency department overcrowding. Med J Aust. 2006 Mar 6;184(5):213-6. doi: 10.5694/j.1326-5377.2006.tb00204.x. PMID 16515430
- [Background] Kwong RY, Schussheim AE, Rekhraj S, Aletras AH, Geller N, Davis J, Christian TF, Balaban RS, Arai AE. Detecting acute coronary syndrome in the emergency department with cardiac magnetic resonance imaging. Circulation. 2003 Feb 4;107(4):531-7. doi: 10.1161/01.cir.0000047527.11221.29. PMID 12566362
- [Background] Ross AM, Gibbons RJ, Stone GW, Kloner RA, Alexander RW; AMISTAD-II Investigators. A randomized, double-blinded, placebo-controlled multicenter trial of adenosine as an adjunct to reperfusion in the treatment of acute myocardial infarction (AMISTAD-II). J Am Coll Cardiol. 2005 Jun 7;45(11):1775-80. doi: 10.1016/j.jacc.2005.02.061. PMID 15936605
- [Background] Mahaffey KW, Puma JA, Barbagelata NA, DiCarli MF, Leesar MA, Browne KF, Eisenberg PR, Bolli R, Casas AC, Molina-Viamonte V, Orlandi C, Blevins R, Gibbons RJ, Califf RM, Granger CB. Adenosine as an adjunct to thrombolytic therapy for acute myocardial infarction: results of a multicenter, randomized, placebo-controlled trial: the Acute Myocardial Infarction STudy of ADenosine (AMISTAD) trial. J Am Coll Cardiol. 1999 Nov 15;34(6):1711-20. doi: 10.1016/s0735-1097(99)00418-0. PMID 10577561
- [Background] Desmet W, Bogaert J, Dubois C, Sinnaeve P, Adriaenssens T, Pappas C, Ganame J, Dymarkowski S, Janssens S, Belmans A, Van de Werf F. High-dose intracoronary adenosine for myocardial salvage in patients with acute ST-segment elevation myocardial infarction. Eur Heart J. 2011 Apr;32(7):867-77. doi: 10.1093/eurheartj/ehq492. Epub 2010 Dec 31. PMID 21196444
- [Background] Thygesen K, Alpert JS, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Redefinition of Myocardial Infarction; Jaffe AS, Apple FS, Galvani M, Katus HA, Newby LK, Ravkilde J, Chaitman B, Clemmensen PM, Dellborg M, Hod H, Porela P, Underwood R, Bax JJ, Beller GA, Bonow R, Van der Wall EE, Bassand JP, Wijns W, Ferguson TB, Steg PG, Uretsky BF, Williams DO, Armstrong PW, Antman EM, Fox KA, Hamm CW, Ohman EM, Simoons ML, Poole-Wilson PA, Gurfinkel EP, Lopez-Sendon JL, Pais P, Mendis S, Zhu JR, Wallentin LC, Fernandez-Aviles F, Fox KM, Parkhomenko AN, Priori SG, Tendera M, Voipio-Pulkki LM, Vahanian A, Camm AJ, De Caterina R, Dean V, Dickstein K, Filippatos G, Funck-Brentano C, Hellemans I, Kristensen SD, McGregor K, Sechtem U, Silber S, Tendera M, Widimsky P, Zamorano JL, Morais J, Brener S, Harrington R, Morrow D, Lim M, Martinez-Rios MA, Steinhubl S, Levine GN, Gibler WB, Goff D, Tubaro M, Dudek D, Al-Attar N. Universal definition of myocardial infarction. Circulation. 2007 Nov 27;116(22):2634-53. doi: 10.1161/CIRCULATIONAHA.107.187397. Epub 2007 Oct 19. No abstract available. PMID 17951284
- [Background] Thygesen K, Alpert JS, Jaffe AS, Simoons ML, Chaitman BR, White HD; Joint ESC/ACCF/AHA/WHF Task Force for the Universal Definition of Myocardial Infarction; Katus HA, Lindahl B, Morrow DA, Clemmensen PM, Johanson P, Hod H, Underwood R, Bax JJ, Bonow RO, Pinto F, Gibbons RJ, Fox KA, Atar D, Newby LK, Galvani M, Hamm CW, Uretsky BF, Steg PG, Wijns W, Bassand JP, Menasche P, Ravkilde J, Ohman EM, Antman EM, Wallentin LC, Armstrong PW, Simoons ML, Januzzi JL, Nieminen MS, Gheorghiade M, Filippatos G, Luepker RV, Fortmann SP, Rosamond WD, Levy D, Wood D, Smith SC, Hu D, Lopez-Sendon JL, Robertson RM, Weaver D, Tendera M, Bove AA, Parkhomenko AN, Vasilieva EJ, Mendis S. Third universal definition of myocardial infarction. Circulation. 2012 Oct 16;126(16):2020-35. doi: 10.1161/CIR.0b013e31826e1058. Epub 2012 Aug 24. No abstract available. PMID 22923432
- [Background] http://www.accordtrial.org/public/documents/Protocol%20All%20Chapters.pdf Accessed 12/12/2011.
- [Background] Puskas JD, Williams WH, Mahoney EM, Huber PR, Block PC, Duke PG, Staples JR, Glas KE, Marshall JJ, Leimbach ME, McCall SA, Petersen RJ, Bailey DE, Weintraub WS, Guyton RA. Off-pump vs conventional coronary artery bypass grafting: early and 1-year graft patency, cost, and quality-of-life outcomes: a randomized trial. JAMA. 2004 Apr 21;291(15):1841-9. doi: 10.1001/jama.291.15.1841. PMID 15100202
- [Background] Vashi AA, Fox JP, Carr BG, D'Onofrio G, Pines JM, Ross JS, Gross CP. Use of hospital-based acute care among patients recently discharged from the hospital. JAMA. 2013 Jan 23;309(4):364-71. doi: 10.1001/jama.2012.216219. PMID 23340638
- [Background] Therneau TM, Grambsch PM, Fleming TR. Martingale-based residuals for survival models 10.1093/biomet/77.1.147. Biometrika 1990;77:147-60.
- [Background] Andersen PK, Gill RD. Cox's Regression Model for Counting Processes: A Large Sample Study. The Annals of Statistics 1982;10:1100-20.
- [Background] Wei LJ, Lin DY, Weissfeld L. Regression Analysis of Multivariate Incomplete Failure Time Data by Modeling Marginal Distributions. Journal of the American Statistical Association 1989;84:1065-73.
- [Background] Prentice RL, Williams BJ, Peterson AV. On the Regression Analysis of Multivariate Failure Time Data. Biometrika 1981;68:373-9.
- [Background] Wong DTL, Das R, Leung MC, et al. Safety of Adenosine Stress Cardiac MRI (AS-CMR) Early after Acute ST Elevation Myocardial Infarction (STEMI) Post-primary Angioplasty. Heart, Lung and Circulation Abstracts for the Cardiac Society of Australia and New Zealand Annual Scientific Meeting and the International Society for Heart Research, Australasian Section, Annual Scientific Meeting 2009;18:S51.
- [Background] Geleijnse ML, Fioretti PM, Roelandt JR. Methodology, feasibility, safety and diagnostic accuracy of dobutamine stress echocardiography. J Am Coll Cardiol. 1997 Sep;30(3):595-606. doi: 10.1016/s0735-1097(97)00206-4. PMID 9283514
- [Background] Noto TJ Jr, Johnson LW, Krone R, Weaver WF, Clark DA, Kramer JR Jr, Vetrovec GW. Cardiac catheterization 1990: a report of the Registry of the Society for Cardiac Angiography and Interventions (SCA&I). Cathet Cardiovasc Diagn. 1991 Oct;24(2):75-83. doi: 10.1002/ccd.1810240202. PMID 1742788
- [Background] Wyman RM, Safian RD, Portway V, Skillman JJ, McKay RG, Baim DS. Current complications of diagnostic and therapeutic cardiac catheterization. J Am Coll Cardiol. 1988 Dec;12(6):1400-6. doi: 10.1016/s0735-1097(88)80002-0. PMID 2973480
- [Background] Nagel E, Lehmkuhl HB, Bocksch W, Klein C, Vogel U, Frantz E, Ellmer A, Dreysse S, Fleck E. Noninvasive diagnosis of ischemia-induced wall motion abnormalities with the use of high-dose dobutamine stress MRI: comparison with dobutamine stress echocardiography. Circulation. 1999 Feb 16;99(6):763-70. doi: 10.1161/01.cir.99.6.763. PMID 9989961
- [Background] Kwong RY, Arai AE. Detecting patients with acute coronary syndrome in the chest pain center of the emergency department with cardiac magnetic resonance imaging. Crit Pathw Cardiol. 2004 Mar;3(1):25-31. doi: 10.1097/01.hpc.0000116584.57152.06. PMID 18340135
- [Background] Ingkanisorn WP, Kwong RY, Bohme NS, Geller NL, Rhoads KL, Dyke CK, Paterson DI, Syed MA, Aletras AH, Arai AE. Prognosis of negative adenosine stress magnetic resonance in patients presenting to an emergency department with chest pain. J Am Coll Cardiol. 2006 Apr 4;47(7):1427-32. doi: 10.1016/j.jacc.2005.11.059. Epub 2006 Mar 20. PMID 16580532
- [Background] Hundley WG, Morgan TM, Neagle CM, Hamilton CA, Rerkpattanapipat P, Link KM. Magnetic resonance imaging determination of cardiac prognosis. Circulation. 2002 Oct 29;106(18):2328-33. doi: 10.1161/01.cir.0000036017.46437.02. PMID 12403662
- [Background] Korosoglou G, Elhmidi Y, Steen H, Schellberg D, Riedle N, Ahrens J, Lehrke S, Merten C, Lossnitzer D, Radeleff J, Zugck C, Giannitsis E, Katus HA. Prognostic value of high-dose dobutamine stress magnetic resonance imaging in 1,493 consecutive patients: assessment of myocardial wall motion and perfusion. J Am Coll Cardiol. 2010 Oct 5;56(15):1225-34. doi: 10.1016/j.jacc.2010.06.020. PMID 20883929
- [Derived] Miller CD, Mahler SA, Snavely AC, Raman SV, Caterino JM, Clark CL, Jones AE, Hall ME, Koehler LE, Lovato JF, Hiestand BC, Stopyra JP, Park CJ, Vasu S, Kutcher MA, Hundley WG. Cardiac Magnetic Resonance Imaging Versus Invasive-Based Strategies in Patients With Chest Pain and Detectable to Mildly Elevated Serum Troponin: A Randomized Clinical Trial. Circ Cardiovasc Imaging. 2023 Jun;16(6):e015063. doi: 10.1161/CIRCIMAGING.122.015063. Epub 2023 Jun 20. PMID 37339173
- See also: Wake Forest Baptist Medical Center — http://www.wakehealth.edu

DOCUMENTS (1):
  • Informed Consent Form (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/52/NCT01931852/ICF_000.pdf